CLINICAL TRIAL: NCT01245543
Title: Open-label, Phase 1 Trial to Evaluate the Safety and Pharmacokinetic Parameters of a 2-day Pulse of Intravenous (IV) AC480 (AC480IV) Administered as Monotherapy and in Combination With Docetaxel in Patients With Advanced Solid Tumors
Brief Title: Safety Study for Intravenous (IV) AC480 (AC480IV) to Treat Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Clinical investigations have been discontinued and transfer to BMS 3/24/2015
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC480IV-001
Record Dates: First submitted 2010-11-17; First posted 2010-11-22 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Docetaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AC480IV (Experimental): Dose range finding study
  Interventions: Drug: Docetaxel
- Docetaxel (Experimental): Dose range finding study in subjects with solid tumors
  Interventions: Drug: AC480IV

INTERVENTIONS:
Drug: AC480IV — AC480IV will be administered as an infusion using a dose escalation design.
  Other Names: AC480IV•Esylate
  Arms: Docetaxel
Drug: Docetaxel — Docetaxel will be administered intravenously, initially as monotherapy and subsequently in combination with docetaxel immediately following AC480IV administration.
  Other Names: Taxol
  Arms: AC480IV

SUMMARY:
AC480IV will be administered as a monotherapy and then in combination with docetaxel in patients with locally advanced or metastatic solid tumors for whom there are no standard or curative therapies available. It is designed to evaluate the safety and pharmacokinetic parameters of AC480IV as monotherapy and also in combination with docetaxel under the conditions of the study.

DETAILED DESCRIPTION:
A Phase I study to determine safety and tolerability of AC480IV with and without Docetaxel in subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥18 years
2. Provide written informed consent
3. Has histological diagnosis of a primary solid tumor malignancy that meets study criteria
4. Has measurable disease (or evaluable if not in MTD expansion cohort) via computed tomography (CT) or magnetic resonance imaging (MRI) scans with or without non-measurable tumors (a lesion in a previously irradiated area is eligible to be considered as measurable disease as long as there is objective evidence of progression of that lesion prior to enrollment)
5. Less than 4 prior systemic cancer therapies (with the exception of hormonal agents), including experimental agents, prior HER-family TKI therapies, and prior docetaxel and other taxane therapy; there are no limits to the number of prior therapies for Part 1
6. Women of childbearing potential (WOCBP) must be using an adequate method of contraception.
7. WOCBP must have a negative serum or urine pregnancy test (sensitivity ≤ 25IU human chorionic gonadotropin [hCG]/L) within 72 hours prior to the start of study drug administration
8. Has an ECOG performance status of 0 or 1
9. Has a life expectancy >3 months
10. Has adequate organ function as determined by laboratory tests

Exclusion Criteria:

1. Patient is currently receiving or has received within the last month prior to Cycle 1 Day 1 (6 weeks for nitrosoureas, mitomycin-C, and liposomal doxorubicin) other chemotherapeutic, hormonal, or investigational anti-cancer agents with the exception of gonadal suppression agents and bisphosphonates for osteoporosis and skeletal metastases which may be continued while on study
2. Patient has received other chemotherapeutic, hormonal, or investigational anti cancer agents that are outside of the timeframe described above and thus would be allowed in the study, but has toxicity that is unresolved (i.e., toxicity has resolved to Grade ≤ 1 or is deemed irreversible)
3. Current or anticipated need for drugs that are known cytochrome P450 isozyme CYP3A4 or CYP2C8 inducers or inhibitors; only exception is oral glucocorticoids, which are a required premedication for docetaxel
4. Patient received previous treatment with oral AC480
5. Patient using herbal and dietary supplements that may interact with CYP3A4
6. Patient received radiation therapy or major surgery within one month of Cycle 1 Day 1
7. Patient has evidence of clinically unstable brain metastases (controlled and stable brain metastasis must be previously treated and asymptomatic)
8. Patient has uncontrolled or significant cardiovascular disease, including:

   * A myocardial infarction within 6 months prior to study entry;
   * Uncontrolled angina within 6 months prior to study entry;
   * History of congestive heart failure (CHF) New York Heart Association (NYHA) class 3 or 4;
   * LVEF that is ≤50% (or ≥ institutional lower limit of normal);
   * Heart rate <50 beats per minute;
   * Diagnosed or suspected congenital long QT syndrome;
   * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes [TdP]);
   * Prolonged corrected interval between the Q wave and T wave (QTc) by Fridericia's correction factor (QTcF) interval on pre-entry ECG ≥450 ms (average of 3 ECG readings done in triplicate);
   * Any history of second or third degree heart block;
   * Uncontrolled hypertension;
   * Obligate need for a cardiac pacemaker;
   * Complete left bundle branch block;
   * Atrial fibrillation; and
   * Abnormal baseline Troponin-I.
9. Patient is using drugs (or has medical conditions) that are generally accepted to have a risk of causing torsades de pointes (TdP) patients who have discontinued any of these medications must have a wash-out period of at least 5 days or 5 half-lives of the drug (whichever is greater) prior to the first dose of AC480IV
10. Patient is in need of anticoagulation therapy except for low-dose heparin or low-dose coumadin for maintenance of patency of central venous access or prevention of deep vein thrombosis (DVT)
11. Women who are pregnant or breastfeeding
12. Male or female patients who are sexually active and unwilling to take contraceptive measures for the duration of the treatments and for 3 months following discontinuation of AC480IV
13. Patient with serious uncontrolled concurrent medical illness including but not limited to ongoing or active infection, and "currently active" second malignancies other than non-melanoma skin cancers
14. Patient with psychiatric illness or social situations that would limit compliance with treatment or adequate informed consent
15. Patient has pre-existing peripheral neuropathy Grade >1
16. Patient has prior hypersensitivity reaction or intolerance to docetaxel or other drugs formulated with polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability, including the dose limiting toxicity (DLT) and the maximum tolerated dose (MTD), of a 2-day pulse of AC480IV both as monotherapy and in combination with docetaxel in patients with advanced solid tumor malignancies. | 18 months
  The primary outcome of the study will be safety and tolerability of the study treatment as measured by physical examinations, adverse events, clinical chemistry evaluations, ECG assessments and the report of dose-limiting toxicity as outlined in the protocol.

SECONDARY OUTCOMES:
Determine the pharmacokinetic (PK) parameters (Cl, Vd, Cmax, Clast, AUClast, AUCinf, t1/2, etc.) of AC480IV and docetaxel as monotherapy and in combination. | Measured at specified timepoints during 1st and/or 2nd cycles of treatment.
  This study is designed to evaluate the safety and PK parameters of AC480IV as monotherapy and also in combination with docetaxel.
Determine any preliminary evidence of efficacy of AC480IV as monotherapy or in combination with docetaxel by assessing tumor response and time to disease progression. | 18 months
  Efficacy assessments will be completed within 7 days after the end of Cycle 3 and then every 3 cycles thereafter. Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) will be used to assess radiographic response.
Evaluate HER profile and Ras mutation status in patients' tumors | Measured in specified dosing cohorts at various timepoints during 1st and/or 2nd cycles of treatment.
  If possible, patients with tumors known to express HER receptors, such as head and neck, lung adenocarcinoma, upper GI/esophageal, and breast cancers will be included.
Evaluate whether AC480IV has anti-metabolic activity in the tumor microenvironment. | Measured in specified dosing cohorts at various timepoints during Part 1 of this study.
  Tumor metabolism will be assessed by comparing pre-dose and postdose assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Gammon, MB BS, MRCP, Study Director — Interim Chief Medical Officer / Ambit Biosciences Corporation
Locations (2):
- United States (2):
  - University of California San Francisco (UCSF), San Francisco, California
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas